CLINICAL TRIAL: NCT03959059
Title: Percutaneous Kyphoplasty Assisted With/Without Mixed Reality Technology in Treatment of OVCF With IVC: a Prospective Study
Brief Title: PKP Assisted With MR Technology in OVCF With IVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20160122-47
Record Dates: First submitted 2019-05-10; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Orthopedic Disorder of Spine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKP of traditional procedure (Experimental): traditional method of PKP
  Interventions: Device: Mixed Reality technology

INTERVENTIONS:
Device: Mixed Reality technology — combine image with real body

SUMMARY:
To prospectively assess the outcome of PKP assisted with and without MR technology in treatment of OVCF with IVC.

DETAILED DESCRIPTION:
The study is to prospectively assess the outcome of PKP assisted with and without MR technology in treatment of OVCF with IVC. Forty cases of OVCF with IVC undergoing PKP were randomized into a MR technology assisted group (group A) and a traditional C-arm fluoroscopy group (group B). Both groups were performed PKP and evaluated by VAS scores, ODI scores, radiological evidence of vertebral body height and kyphotic angle(KA) at pre-operation and post-operation. The volume of injected cement and Operation time was recorded. And whether cement touching both endplates or not(non-PMMA-endplates-contact, NPEC) in radiological evidence were also recorded postoperatively. The clinical outcomes and complications were evaluated afterwards. All patients received 10 to 14 months' follow-up, with an average of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Single level OVCF in the thoracic and lumbar levels (T10-L4), suffering with severe back pain.;
* OVCF without damaged vertebral posterior wall and nerve lesion;
* The patient was over 50 years old and , the diagnosis of osteopenia or osteoporosis was confirmed by bone densitometry ;
* All patients underwent（received） plain radiography, computed tomography (CT) and MRI before surgery, and with IVC presented in MRI.

Exclusion Criteria:

-

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 1 year
  visual analog scale(0-10 scores) is for pain, 0 represent no pain, 10 score represent the severe pain.
Oswestry Disability Index | 1 year
  Oswestry Disability Index is for movement function, Questionnaire examines perceived level of disability in everyday activities of daily living. The ODI score (index) is calculated as: For example: If all 10 sections are completed, the score is calculated as follows: if 16 (total scored) out of 50 (total possible score) x 100 = 32%; If one section is missed (or not applicable), the score is calculated: If 16 (total scored) / 45 (total possible score) x 100 = 35.5%.
Vertebral height | 1 year
  Vertebral height in X-ray is for recontruction of the vertebra.
Kyphotic angle | 1 year
  kyphotic angle in X-ray is also for recontruction of the vertebra.

CONTACTS AND LOCATIONS:
Locations (1):
- Mixed Reality, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wei P, Yao Q, Xu Y, Zhang H, Gu Y, Wang L. Percutaneous kyphoplasty assisted with/without mixed reality technology in treatment of OVCF with IVC: a prospective study. J Orthop Surg Res. 2019 Aug 8;14(1):255. doi: 10.1186/s13018-019-1303-x. PMID 31395071